CLINICAL TRIAL: NCT02655276
Title: Effects of Sublingual Microencapsulated Glycine on Attentional Difficulties and Hyperactivity in Prepuberal Children - A Placebo-controlled, Double-blind, Randomized, Cross-over Study
Brief Title: Sublingual Glycine vs. Placebo on Attentional Difficulties and Hyperactivity in Prepuberal Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eberhard Schulz (Other)
Collaborators: Biotiki (Unknown)
Responsible Party: Sponsor-Investigator, Eberhard Schulz, Prof. Dr., University Hospital Freiburg
Organization: University Hospital Freiburg (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Classroom FR03
Record Dates: First submitted 2016-01-08; First posted 2016-01-14 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Motor Activity; Attention Deficit; Stress, Psychological
Keywords: microencapsulated glycine; attentional performance; motoric activity; hyperactivity
MeSH Terms: conditions — Motor Activity; Attention Deficit Disorder with Hyperactivity; Stress, Psychological; Spasm

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 100 mg microencapsulated Glycine and then Placebo tablets (Experimental): 100 mg microencapsulated Glycine (Bidicin® from Biotiki® ) t.i.d. for the first three weeks and then Placebo t.i.d. from Biotiki® for the second three weeks.
  Interventions: Other: microencapsulated Glycine; Other: Placebo tablets
- Placebo tablets and then 100 mg microencapsulated Glycine (Experimental): Placebo t.i.d. from Biotiki® for the first three weeks and then 100 mg microencapsulated Glycine (Bidicin® from Biotiki® ) t.i.d. for the second three weeks.
  Interventions: Other: microencapsulated Glycine; Other: Placebo tablets

INTERVENTIONS:
Other: microencapsulated Glycine — 100 mg microencapsulated Glycine (Bidicin® from Biotiki® ) t.i.d.
Other: Placebo tablets — Placebo t.i.d. from Biotiki® in a crossover-design.

SUMMARY:
This study is designed to investigate effects on attentional performance and motoric activity of 100 mg microencapsulated glycine (Bidicin® from Biotiki®) compared to placebo after treatment with t.i.d. sublingual doses over 3 weeks each.

The primary objective of the study is to determine the effects on attentional performance and motoric activity of 100 mg microencapsulated Glycine (Bidicin® from Biotiki® ) compared to placebo after treatment with t.i.d. sublingual doses over 3 weeks each in children with low attentional performance and high motoric activity.

A number of 30 prepuberal boys and girls aged 6 - 14 years with low attentional performance and high motoric activity will be enrolled in this study. The prepuberal status will be determined by Tanner stages ≤ 3.

DETAILED DESCRIPTION:
Trial Design:

This study has a double-blind, randomized, two-period, cross-over design. The study population will be randomized equally to the sequence 1 (first 3 weeks microencapsulated Glycine, second 3 weeks placebo) or sequence 2 (first 3 weeks placebo, second 3 weeks microencapsulated Glycine). Study Agent/Placebo - Dosage and Route of Administration:

Study Agent/Placebo will first be dispensed at Visit 2 (day 0). Treatment assignments will be made in accordance with the randomization. At each visit (Visit 2 and Visit 3), subjects will receive two blisters for the 3 following weeks. Only qualified personnel may dispense study Agent/Placebo.

Investigational and reference treatment:

100 mg microencapsulated Glycine (Bidicin® from Biotiki® ) Placebo from Biotiki®

Study design:

This study will employ a double blind, randomized, placebo-controlled cross-over design. SKAMP raters and teachers will be blinded concerning the study Agent/Placebo.

Planned Study Time Schedule:

The study ends 10 weeks after enrollment of the last patient (total study end). Study duration for each patient is between 7 and 10 weeks (from inclusion) until the last visit (close-out visit).

Statistics:

Sample size calculation is based on the primary endpoint "mean of the SKAMP Combined score over all time points in the classroom setting". The study should have sufficient power to detect a difference between treatments if a moderate effect size (corresponding to Cohen's d=0.5) were present in parallel-group study in two independent patient groups. Assuming a correlation between measurements in the same patient of 0.6, this translates into an effect size of 0.56 in a cross-over trial comparing within patient measurements. With this effect size, 27 patients have to be included in the study, to achieve a power of 0.8 at a two-sided significance level of alpha=0.05. To account for a small number of drop-outs, 30 patients have to be randomized.

Data analysis: The trial will be analyzed according to the intention-to-treat principle. Efficacy measures will be evaluated by linear mixed models for repeated measurements.

Safety analyses will be performed for subjects who received at least one dose of microencapsulated Glycine/ placebo. Incidences of adverse events and of serious adverse events will be calculated.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all of the following inclusion criteria will be eligible for enrollment in the study:

1. Male and female subjects aged 6-14 years with Tanner stages 0 to 3 and attentional and/or hyperactivity problems.
2. Subjects with parents or a legal guardian, who will give written informed consent for the child to participate in the study. Additionally, assent to participate must be obtained from all children entering the study if the child is able to judge the nature, the meaning and the significance of the trial. Assent will be documented by the child´s signature on the consent form.
3. Health Status: Subjects must not have clinically significant diseases or clinically significant abnormal laboratory values as assessed during medical history and physical exam.
4. Subjects meeting minimum intelligence requirements: In the opinion of the investigator the subject must generally be functioning at age-appropriate levels academically, which should take into account any prior cognitive or academic testing (basic knowledge of reading, writing and calculating).
5. Subject has an ADHD-RS-IV total score ≥18.
6. Subjects already receiving behavioral therapies for HKS/ADHD or oppositional defiant disorder may continue to do sor during the course of the trial.

Exclusion Criteria:

1. subjects with psychiatric disorders requiring current pharmacological treatment (e.g. major depression, psychosis)
2. Subjects with psychiatric or somatic conditions that may contraindicate the trial or confound efficacy or safety assessments.
3. Subjects with a history of drug abuse or current use of recreational drugs.
4. History of hypersensitivity to microencapsulated Glycine or placebo.
5. Subjects who are judged by the investigator as likely to be non-compliant with study procedures.
6. Use of any investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer.
7. History of malignancy of any organ system, treated or untreated, within the past 5 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
SKAMP-Combined rating scale in the classroom setting | 3 weeks
  SKAMP-Combined rating performed at 25 minutes before and 0:50 h, 1,55 h, 2:50 h, 4:05 h, 5:50 h, 7:40 h and 8:35 h after first microencapsulated Glycine/ placebo intake in a laboratory classroom setting after a 3 week treatment period. The primary efficacy endpoint is the mean of the SKAMP-Combined score over all time points in the classroom setting.

SECONDARY OUTCOMES:
SKAMP-Attention subscale | 3 weeks
  SKAMP- Attention subscale rating performed at 25 minutes before and 0:50 h, 1,55 h, 2:50 h, 4:05 h, 5:50 h, 7:40 h and 8:35 h after first microencapsulated Glycine/ placebo intake in a laboratory classroom setting after a 3 week treatment period. The secondary efficacy endpoint is the mean of the SKAMP- Attention subscale score over all time points in the classroom setting.
SKAMP-Deportment subscale | 3 weeks
  SKAMP- Deportment subscale rating performed at 25 minutes before and 0:50 h, 1,55 h, 2:50 h, 4:05 h, 5:50 h, 7:40 h and 8:35 h after first microencapsulated Glycine/ placebo intake in a laboratory classroom setting after a 3 week treatment period. The secondary efficacy endpoint is the mean of the SKAMP- Deportment subscale score over all time points in the classroom setting.
Child Behaviour Checklist (CBCL) | 3 weeks
  The assessment of the child behaviour scale (CBCL) is performed by the primary caregivers due to the last week before the visit of a classroom. The CBCL global score and the CBCL subscores are used for evaluation.
Quality of life scores | 3 weeks
  The instrument provides a QoL total score and several domains of QoL regarding family, school, peers, interests, physical and mental health, and also the impact of the respective disorder. These scores are used for evaluation.
Visual-Analogue-Scale of perceived parental stress | 3 weeks
  The value of the visual-analogue-scale of perceived parental stress is used for evaluation.
Saliva cortisol levels | 3 weeks
  In this study, saliva cortisol samples are collected for determination of the cortisol awakening response (CAR) as well as before and after the supposedly stressful situation of the classroom math test. For the CAR, cortisol will be measured on three consecutive days before Visit 2, 3 and 4 at awakening, 30 minutes after awakening and before bedtime.
  For assessment of cortisol levels under acute stress, cortisol samples will be taken before and after classroom III of Visit 2, as well as before and after classroom III and VI of Visits 3 and 4.
ADHD-Rating scale-IV | 3 weeks
  The ADHD Rating Scale-IV is a reliable and easy-to-administer instrument both for diagnosing ADHD in children and adolescents and for assessing treatment response. Containing 18 items, the scale is linked directly to DSM-IV diagnostic criteria for ADHD.
  Outcome Measure are the summed total score for "Inattention, Hyperactivity and Impulsivity" and the sub-scores for "Inattention" and for "Hyperactivity and Impulsivity".
Adverse Events that are related or not related to treatment | 3 weeks
  All adverse events no matter how intense will be observed by the investigator until resolved or until they can be sufficiently medical explained. All AEs must be described by diagnosis or symptoms, duration, frequency, severity, an assessment of its cause, its relationship to the study Glycine or placebo, whether it influenced the course of the study Glycine or placebo, whether it required specific therapy and its outcome.
  All documented AEs will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Eberhard Schulz, Prof. Dr., Study Director — University Hospital Freiburg
Locations (1):
- University Hospital, Freiburg im Breisgau, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No